CLINICAL TRIAL: NCT04986410
Title: Quantitative Analysis of Functional Computed Tomography (CT) Imaging of Coronary Atherosclerosis
Brief Title: Quantitative Analysis of Functional CT Imaging of Coronary Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016YFC1300302
Record Dates: First submitted 2021-07-11; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: CT myocardial perfusion imaging; SPECT myocardial perfusion imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial Perfusion examination
  Interventions: Diagnostic Test: CCTA, CT-MPI, CT-FFR, SPECT-MPI

INTERVENTIONS:
Diagnostic Test: CCTA, CT-MPI, CT-FFR, SPECT-MPI — Subjects undergo CCTA, CT-MPI, CT-FFR or SPECT-MPI

SUMMARY:
The purpose of this prospective observational study is to evaluate the diagnostic and prognostic performance of a "one-stop" comprehensive coronary artery anatomy and function assessment for CAD.

DETAILED DESCRIPTION:
Coronary CT angiography (CCTA) has become a reliable diagnostic technique to evaluate coronary artery disease (CAD) with high sensitivity and a negative predictive value. However, CCTA provides only anatomic information and tends to overestimate stenosis severity and is limited in its ability to diagnose myocardial ischemia. Undertaking additional CT myocardial perfusion imaging(CT-MPI) and CT-FFR improves specificity and positive predictive value, reducing unnecessary invasive coronary angiography. The purpose of this prospective observational study is to evaluate the diagnostic and prognostic performance of a "one-stop" comprehensive coronary artery anatomy and function assessment for CAD. SPECT myocardial perfusion imaging (SPECT-MPI)and invasively measured fractional flow reserve (FFR) will serve as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Understand the purpose of the trial, voluntarily participate in this study, and have signed an informed consent form.
3. Patients with known or suspected CAD

Exclusion Criteria:

1. Patients with acute coronary syndrome.
2. Severe cardiac dysfunction (LVEF ≤ 0.3).
3. Cardiomyopathy with non-coronary causes such as hypertrophic cardiomyopathy, dilated cardiomyopathy, alcoholic cardiomyopathy, and myocardial amyloidosis.
4. Severe cardiac valve disease with more than moderate valvular regurgitation and/or valvular stenosis.
5. Severe hepatic and renal dysfunction (ALT ≥ 3 Upper Limit of Normal, Cr> 134μ/mol/L (2mg/dl) or estimated Glomerular Filtration Rate<45ml/min/1.73m2).
6. Severe arrhythmias (persistent atrial fibrillation, second-degree or third-degree atrioventricular block, etc.)
7. Malignancy or other pathophysiological conditions with an expected survival of less than 1 year
8. Allergic to the drug components involved in this study and those who are intolerant to loading tests
9. Pregnant or lactating women.
10. Mental disorders.
11. Failure to sign the informed consent form.
12. Other conditions that are incompatible with the clinical study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected CAD
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 5 years
  including cardiac death, all-cause death, acute coronary syndrome, readmission for acute coronary syndrome or heart failure, and Revascularization.

SECONDARY OUTCOMES:
Diagnostic performance of CT-MPI | From admission to discharge, up to 1 week
  Diagnostic accuracy, Sensitivity, specificity, negative predictive value(NPV) and positive predictive value(PPV) of CT-perfusion imaging (quantitative and qualitative analysis) to determine the presence/absence of significant coronary artery disease at the subject level when compared with invasive FFR and SPECT-MPI.
Diagnostic performance of CT-FFR | From admission to discharge, up to 1 week
  Diagnostic accuracy, Sensitivity, specificity, negative predictive value(NPV) and positive predictive value(PPV) of CT-FFR to determine the presence/absence of significant coronary artery disease at the subject level when compared with invasive FFR and SPECT-MPI.
Diagnostic performance of CT-MPI | From admission to discharge, up to 1 week
  Diagnostic accuracy, Sensitivity, specificity, negative predictive value(NPV) and positive predictive value(PPV) of CT-perfusion imaging (quantitative and qualitative analysis) to determine the presence/absence of significant coronary artery disease in per-vessel level when compared with invasive FFR and SPECT-MPI.
Diagnostic performance of CT-FFR | From admission to discharge, up to 1 week
  Diagnostic accuracy, Sensitivity, specificity, negative predictive value(NPV) and positive predictive value(PPV) of CT-FFR to determine the presence/absence of significant coronary artery disease in per-vessel level when compared with invasive FFR and SPECT-MPI.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Zhang, Study Chair — Qilu Hospital of Shandong University; Mei Zhang, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No